CLINICAL TRIAL: NCT05252377
Title: Investigation of the Effect of Breathing Exercise on Invasive Pain Associated With Arteriovenous Fistula Cannulation in Hemodialysis Patients.
Brief Title: Breathing Exercise and Invasive Pain at Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Demiroglu Bilim University (Other)
Responsible Party: Principal Investigator, Nurten Ozen, Associate Professor, Istanbul Demiroglu Bilim University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2021-20-02
Record Dates: First submitted 2022-02-14; First posted 2022-02-23 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Pain; Arteriovenous Fistula; Breathing Exercise
MeSH Terms: conditions — Pain; Arteriovenous Fistula | interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Breathing Exercise Group (Experimental): Breathing exercise program; It was prepared by the researchers in accordance with the literature and based on the studies in which breathing exercise was applied to reduce invasive pain experienced during cannulation, blood collection and postoperative pain. Patients will be given an exercise based on rhythmic breathing. The exercise will be started before the cannulation application, the patient will be told to perform the breathing exercise twice, and he will be asked to continue doing the breathing exercise until the cannulation process is completed. The patient will wait by taking five normal breaths between each breathing exercise. The patient will be told that he can count by using his fingers in the steps he is asked to count up to three.
  Interventions: Other: Breathing Exercise
- Control Group (No Intervention): No intervention will be made by the researcher on the patients in this group, and a pain assessment will be made by the nurse in charge of dialysis immediately after the cannulation procedure by the dialysis nurse working in the unit.

INTERVENTIONS:
Other: Breathing Exercise — 1. The patient will be asked to close their eyes
  2. He will be asked to relax his head and neck in a semi-sitting position in bed
  3. The patient will be asked to breathe through the nose for 3 seconds by counting
  4. Then he will be told to hold his breath for 3 seconds
  5. As the last step, he will be asked to breathe out again in 3 seconds.
  Arms: Breathing Exercise Group

SUMMARY:
Non-pharmacological approaches applied in the prevention of invasive pain due to cannulation in patients treated with arteriovenous fistula and hemodialysis; It is also a cost-effective method that prevents the patient from feeling pain from the application. Breathing exercises are a method that can be easily applied before the cannulation procedure. Although it is seen that there are limited number of studies on the subject in the literature, it was observed that the duration of breathing exercise application was short (two weeks) in one study and the duration was not specified in the other.

DETAILED DESCRIPTION:
An average of 312 cannulations per year is performed in a patient who is treated for chronic hemodialysis and has arteriovenous fistula. Patients state that they experience moderate to severe pain at a rate of 57-60.9% when accessing the arteriovenous. In cases where access to the fistula cannot be achieved at one time, patients may experience pain due to; patients experience non-compliance with dialysis treatment and their quality of life is adversely affected. This situation causes an increase in the mortality rate, especially with cardiovascular and respiratory system complications. In recent years, breathing exercise, which is one of the methods of distraction, has been used to reduce the invasive pain experienced during blood collection and cannulation procedures. By increasing lung ventilation with breathing, the amount of oxygen entering the body is maximized, and this causes relaxation in the patient. This relaxation also causes the person to relax and reduce the pain they will feel. Although studies have found that breathing exercise is effective in reducing invasive pain; No information was given about the exercise method and duration. Although in practice, holding the patient's breath during venipuncture and performing the cannulation procedure while giving it is a method frequently applied by the nurse, no study with high evidence supporting the situation has been found in the literature.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis treatment with arteriovenous for at least 3 months
* Hemodialysis treatment is applied for 3 days and 4 hours a week.
* Between the ages of 18-65
* Pain score ≥ 2 as assessed by Visual Analogue Scale during cannulation of the arteriovenous fistula
* Absence of advanced heart failure, asthma and chronic obstructive pulmonary disease
* Able to communicate in Turkish
* Not having any psychiatric disorder that prevents communication
* Agreeing to participate in the research

Exclusion Criteria:

* Inability to do breathing exercises properly
* Presence of infection, edema and scar tissue in the area where the arteriovenous fistula is located
* Using pain medication before hemodialysis treatment
* Two or more cannulation attempts for arteriovenous fistula in the same session
* Presence of neuropathy and peripheral vascular disease
* Pregnancy
* Withdrawal from the study at any stage of the research

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-01-05 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-05-01 (Actual)

PRIMARY OUTCOMES:
Change From Baseline Invasive Pain at 12 Dialysis Session | At the end of the every dialysis session during one month (3 hemodialysis sessions are done every week)]
  It will be assessed total 12 times at the end of the dialysis session with Visual Analogue. Pain intensity measured on a Visual Analog Scale with scores ranging from 0 - 10. Pain increases as the score increases. The high point describes bad outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Demiroglu Bilim University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alzaatreh MY, Abdalrahim MS. Management Strategies for Pain Associated with Arteriovenous Fistula Cannulation: An Integrative Literature Review. Hemodial Int. 2020 Jan;24(1):3-11. doi: 10.1111/hdi.12803. Epub 2019 Dec 3. PMID 31797508
- [Background] Aitken E, McLellan A, Glen J, Serpell M, Mactier R, Clancy M. Pain resulting from arteriovenous fistulae: prevalence and impact. Clin Nephrol. 2013 Nov;80(5):328-33. doi: 10.5414/CN107917. PMID 23743153
- [Background] Crespo Montero R, Rivero Arellano F, Contreras Abad MD, Martinez Gomez A, Fuentes Galan MI. Pain degree and skin damage during arterio-venous fistula puncture. EDTNA ERCA J. 2004 Oct-Dec;30(4):208-12. doi: 10.1111/j.1755-6686.2004.tb00369.x. PMID 15835412